CLINICAL TRIAL: NCT01713309
Title: Heparin Binding Protein in Patients With Acute Respiratory Failure Treated With Granulocyte Colony-stimulating Factor (Filgrastim)
Brief Title: Heparin Binding Protein in Patients With Acute Respiratory Failure Treated With GCSF (Filgrastim)
Acronym: HBP-Neupogen
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: The Swedish Research Council (Other Government)
Responsible Party: Principal Investigator, Kirsi-Maija Kaukonen, MD, PhD, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HBP01
Record Dates: First submitted 2012-10-14; First posted 2012-10-24 (Estimated); Last update posted 2012-10-29 (Estimated); Status verified 2012-10

CONDITIONS: Acute Respiratory Failure; Critically Ill
Keywords: Filgrastim; G-CSF; Heparin-binding protein; critically ill; acute respiratory failure
MeSH Terms: conditions — Critical Illness | interventions — Filgrastim

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Filgrastim (Active Comparator): Filgrastim 300 microgr/day subcutaneously for 7 days
  Interventions: Drug: Filgrastim
- NaCl 0.9% (Placebo Comparator): Corresponding placebo once daily, subcutaneously for 7 days

INTERVENTIONS:
Drug: Filgrastim — Filgrastim 300 ug daily for 7 days, subcutaneously.
  Other Names: Neupogen
  Arms: Filgrastim

SUMMARY:
This is a study of plasma HBP -levels of a previously published trial of G-CSF in critically ill patients (Pettila et al. Critical Care Medicine 2000). The original study was a prospective, randomised, double-blind, placebo-controlled trial of filgrastim in patients with acute respiratory failure requiring intubation. In this substudy, the investigators evaluated the effect of filgrastim on HBP -concentrations in critically ill patients.

ELIGIBILITY:
Criteria for original study. For the substudy, all these patients were included.

Inclusion Criteria:

* Age > 18 years
* Admitted to the ICU no longer than 12 hrs before study entry
* Intubated because of ventilation insufficiency no longer than 48 hrs before study entry
* Clinically expected stay in the ICU > 48 hrs
* Informed consent

Exclusion Criteria:

* Pregnant or nursing
* Total leukocyte count of > 50,000/mm3
* Administration of filgrastim, sargramostim, or other biological response modifiers within 7 days before study entry
* Known hypersensitivity or allergic reaction to Escherichia coli-derived products
* Participation in another drug study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 1996-01; Primary Completion 1998-06 (Actual); Study Completion 1998-09 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | up to 28 days
  the number of patients developing ARDS, disseminated intravascular coagulation or acute renal failure during days 1-28, and changes in MOD score during days 1-7.

SECONDARY OUTCOMES:
follow up measures | Up to day 90
  frequency of nosocomial infections, length of mechanical ventilatory support, length of stay in the ICU, 28-day mortality rate, 90-day mortality rate, and laboratory values for neutrophil count

OTHER OUTCOMES:
inflammatory mediators | up to day 7
  cytokines, IL-6, TNF, phospolipase A2 and BPIP (=bacterial permeability increasing protein)

CONTACTS AND LOCATIONS:
Overall Officials: Ville Pettila, MD, PhD, Study Director — Helsinki University Central Hospital; Kirsi-Maija Kaukonen, MD, PhD, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Helsinki University Central Hospital, Helsinki, Finland

REFERENCES:
- [Result] Pettila V, Takkunen O, Varpula T, Markkola A, Porkka K, Valtonen V. Safety of granulocyte colony-stimulating factor (filgrastim) in intubated patients in the intensive care unit: interim analysis of a prospective, placebo-controlled, double-blind study. Crit Care Med. 2000 Nov;28(11):3620-5. doi: 10.1097/00003246-200011000-00011. PMID 11098963
- [Result] Takala A, Pettila V, Takkunen O, Rintala E, Kautiainen H, Repo H. Granulocyte colony-stimulating factor therapy and systemic inflammation in critically ill patients. Inflamm Res. 2005 Apr;54(4):180-5. doi: 10.1007/s00011-005-1340-2. PMID 15883741
- [Derived] Kaukonen KM, Herwald H, Lindbom L, Pettila V. Heparin binding protein in patients with acute respiratory failure treated with granulocyte colony-stimulating factor (filgrastim)--a prospective, placebo-controlled, double-blind study. BMC Infect Dis. 2013 Jan 30;13:51. doi: 10.1186/1471-2334-13-51. PMID 23363492